CLINICAL TRIAL: NCT01112787
Title: A Phase 1, Evaluator-Blinded, Randomized, Vehicle Controlled, Study To Evaluate The Cumulative Irritation Potential Of Topically Applied Tazarotene Foam In Healthy Volunteers
Brief Title: A Study to Evaluate the Irritation Potential of Tazarotene Foam on Skin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 114571
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Acne Vulgaris
Keywords: Healthy Volunteer Subjects
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tazarotene Foam (Experimental): Subjects will be exposed to patches containing Tazarotene Foam 0.1%,
  Interventions: Drug: Tazarotene Foam
- Vehicle Foam (Placebo Comparator): Subjects will be exposed to patches containing Vehicle Foam.
  Interventions: Drug: Vehicle Foam
- Sodium Laural Sulfate (Active Comparator): Subjects will be exposed to patches containing Sodium Laural Sulfate.
  Interventions: Drug: Sodium Laural Sulfate
- Distilled Water (Placebo Comparator): Subjects will be exposed to patches containing Distilled Water.
  Interventions: Drug: Distilled Water

INTERVENTIONS:
Drug: Tazarotene Foam — Tazarotene Foam
  Arms: Tazarotene Foam
Drug: Vehicle Foam — Vehicle Foam
  Arms: Vehicle Foam
Drug: Sodium Laural Sulfate — Sodium Laural Sulfate
  Arms: Sodium Laural Sulfate
Drug: Distilled Water — Distilled Water
  Arms: Distilled Water

SUMMARY:
The purpose of this study is to evaluate the irritation level of tazarotene foam after 21 days of exposure on the skin of healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, single center, evaluator-blinded, randomized, vehicle controlled study to evaluate the potential of tazarotene foam to induce cutaneous irritation using a 21 day cumulative irritation assay in healthy adult volunteers. Approximately 40 healthy male and female volunteer subjects aged 18 to 65 years will be enrolled. All subjects will be exposed to patches containing tazarotene foam, vehicle foam, sodium lauryl sulfate 0.5% (positive control), and distilled water (negative control). Each set of patches will be applied to the same randomized sites once daily for 21 days; patches will be removed after 24 ±1 hours and the patch sites will be evaluated for signs inflammatory skin responses (eg, erythema, edema, papules) and superficial effects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent and Health Information Portability and Accountability Act (HIPAA) authorization before any protocol-specific procedures are performed.
* Male or female aged 18 to 65 years, inclusive, at time of consent.
* Able and willing to complete the study and to comply with all study instructions.
* Possess Fitzpatrick skin types I (always burns easily; never tans), II (always burns easily; tans minimally), III (burns moderately; tans gradually), or IV (rarely burns; tans with ease) that will not interfere with the evaluation of any skin responses .
* Male subjects and their partners must agree to use a medically acceptable method of contraception.
* Additional criteria for women of childbearing potential, defined as one who is biologically capable of becoming pregnant, including perimenopausal women who are less than 2 years from their last menses:

  * A regular menstrual cycle before study entry (as reported by the subject).
  * Negative urine pregnancy test within 2 weeks of the first application of study product.
  * Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception throughout the duration of the study.

Women who are not currently sexually active must agree to use a medically acceptable method of contraception should they become sexually active while participating in the study.

Exclusion Criteria:

* Female who is pregnant, trying to become pregnant, or breast feeding.
* Considered unable or unlikely to attend the necessary visits.
* History of known or suspected intolerance to tazarotene, any of the ingredients of the study products, the hypoallergenic tape, or the cotton patches.
* Participation in any patch test study within 4 weeks of the Day 1 visit.
* Inability to evaluate the skin in and around the potential patch test sites on the back due to sunburns, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality.
* Clinically significant skin diseases that may contraindicate participation or interfere with patch test site evaluations, including psoriasis, eczema, atopic dermatitis, acne, dysplastic nevi, or other skin pathologies, or a history of skin cancer.
* Any major illness within 4 weeks of the Day 1 visit.
* Considered immunocompromised.
* A clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* Clinically relevant history or currently suffering from any disease or condition that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk. This may include respiratory (including chronic asthma requiring repetitive drug interventions), gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders.
* Received any investigational product or procedure within 4 weeks of the Day 1 visit or who is scheduled to receive an investigational product (other than the study product) or procedure during the study.
* Received allergy injections within 1 week of the Day 1 visit, or expects to receive allergy injections during study participation.
* Received immunizations within 4 weeks of the Day 1 visit.
* Used systemic or topical corticosteroids or other immunosuppressive medications within 4 weeks of the Day 1 visit.
* Used topical medications or other products (eg, self tanning products, waxing products, benzoyl peroxide, salicylic acid, or sulfur) in the areas of patch testing within 2 weeks of the Day 1 visit.
* Used antihistamines, selective leukotriene receptor antagonists (eg, montelukast sodium, zafirlukast), or mast cell stabilizers (eg, cromolyn sodium or nedocromil sodium) within 4 weeks of the Day 1 visit.
* Used nonsteroidal anti-inflammatory medications within 2 weeks of the Day 1 visit.
* Currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Participated in a previous study of the same study product.
* Employee of the study center, contract research organization, or Stiefel who is involved in the study, or an immediate family member (eg, partner, offspring, parents, siblings or sibling's offspring) of an employee who is involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-03-26 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2010-04-26 (Actual)

PRIMARY OUTCOMES:
Inflammatory skin responses | 21 days
  Patch sites will be evaluated for signs of inflammatory skin responses (e.g. erythema, edema, papules) and superficial effects.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- HillTop Research Corporation, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114571 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114571?search=study&search_terms=114571#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register